CLINICAL TRIAL: NCT01268397
Title: Unstable Dorsally Displaced Fractures of the Distal Radius in the Elderly. A Randomized Comparison Between Operative Fixation and Plaster Cast Treatment.
Brief Title: Unstable Dorsally Displaced Fractures of the Distal Radius in the Elderly
Acronym: VOCAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Sara Severin Wahlgren, MD, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wilcke-02
Record Dates: First submitted 2010-12-29; First posted 2010-12-30 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2018-04

CONDITIONS: Fracture of the Distal Radius; Wrist Fracture
Keywords: elderly; wrist fracture; fracture of the distal radius; volar plate; plaster cast
MeSH Terms: conditions — Wrist Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORIF (Active Comparator): Open reduction and internal fixation with a volar plate
  Interventions: Procedure: open reduction and internal fixation with a volar plate
- plaster treatment (Active Comparator): Closed reduction and plaster treatment
  Interventions: Procedure: closed reduction and plaster treatment

INTERVENTIONS:
Procedure: open reduction and internal fixation with a volar plate — flexor carpi radialis approach, open reduction, fixed-angle volar plate, plaster cast 2 weeks at the surgeon's discretion
  Other Names: plate: Königsee or Aculoc from Swemac, Sweden
  Arms: ORIF
Procedure: closed reduction and plaster treatment — closed reduction, below elbow plaster cast, semicircular for 5 week
  Arms: plaster treatment

SUMMARY:
The purpose of this study is to examine whether operation and fixation with a metal plate gives better result from the patient's perspective than plaster treatment in elderly patients with a displaced wrist fracture.

DETAILED DESCRIPTION:
We will perform a prospective randomized clinical trial comparing open reduction and internal fixation with a volar plate with closed reduction and plaster treatment in elderly patients with a displaced Colles' fracture in order to test the null hypothesis that the patient-perceived result is equal after conservative or operative treatment. Secondary outcomes are objective physical measurements.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral unstable dislocated dorsally angulated fracture of the distal radius (radial shortening ≥4 mm and/or dorsal angulation ≥20°).

Exclusion Criteria:

* Previous displaced fracture of the distal radius.
* Additional fractures of the upper extremities, an open fracture, terminal disease, patient not fit for surgery, unwilling or unable to co-operate with follow-up (advanced dementia (SPMSQ<5), psychiatric illness, alcohol abuse).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2018-01 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
patient-perceived disability measured by the PRWE and DASH questionnaires | one year after wrist fracture

SECONDARY OUTCOMES:
impairments (grip strength and range of motion compared with the uninjured wrist) | one year after wrist fracture

CONTACTS AND LOCATIONS:
Overall Officials: Per Y Adolphson, MD, PhD, Study Director — Karolinska Institute at Danderyd Hospital
Locations (1):
- Division of Orthopaedics Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sudow H, Severin S, Wilcke M, Saving J, Skoldenberg O, Navarro CM. Non-operative treatment or volar locking plate fixation for dorsally displaced distal radius fractures in patients over 70 years - a three year follow-up of a randomized controlled trial. BMC Musculoskelet Disord. 2022 May 12;23(1):447. doi: 10.1186/s12891-022-05394-7. PMID 35549696